CLINICAL TRIAL: NCT02574507
Title: Behavioral Weight and Symptom Management for Breast Cancer Survivors and Partners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00063328; 1F32CA200091-01 (NIH)
Record Dates: First submitted 2015-10-05; First posted 2015-10-14 (Estimated); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Breast Cancer
Keywords: breast cancer; weight management; couples; symptom management
MeSH Terms: conditions — Breast Neoplasms | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Couples-Based Behavioral Weight and Symptom Management (Experimental): Participants will receive 12 session (6 weekly and 6 biweekly) of a behavioral weight and symptom management intervention.
  Interventions: Behavioral: Couples-Based Behavioral Weight and Symptom Management

INTERVENTIONS:
Behavioral: Couples-Based Behavioral Weight and Symptom Management — Investigators anticipate that the intervention developed in phase I will consist of a total of 12 sessions 90 minutes in length (18 therapy hours) spaced across approximately 5 months. Sessions are spaced to provide participants sufficient time to complete home practice exercises and adequately examine change in weight and maintenance of weight loss. Sessions will be conducted individually for each day. The first 6 sessions will occur weekly and the final 6 sessions will occur biweekly.

SUMMARY:
The objective of the study is to develop and test the feasibility, acceptability, and initial efficacy of a novel couples-based behavioral weight and symptom management intervention for obese breast cancer survivors and their partners. The proposed project consists of two phases. Phase I will include intervention development and refinement. Intervention development will be guided by the research team's prior work, the interdependence model of communal coping and behavior change, and information obtained from couples participating in focus groups. The intervention protocol will then be tested with 5 couples to assist with refinement of intervention content. During phase II, the feasibility, acceptability and initial efficacy of the intervention will be examined. Obese breast cancer survivors in the three years following treatment and their overweight or obese partners will receive 6 weekly and 6 biweekly sessions for a total of 12 sessions spaced across approximately 5 months. The intervention will be provided in a couples-based format where each couple will meet separately with the therapist. Couples will be assessed at pre-, post-, and 3-months post-treatment. Study outcomes will be weight, symptoms (i.e., pain, fatigue, distress), eating behavior, and physical activity. Exploratory outcomes examine biomarkers (i.e., insulin, IL-6, IL-8, TNF-alpha, adiponectin) associated with health outcomes for cancer survivors and their partners. It is hypothesized that the intervention will be feasible (i.e., completed sessions), and participants will find the intervention acceptable as assessed by a measure of treatment acceptability. It is also hypothesized that participants will evidence decreased weight and improvements in symptoms (i.e., pain, fatigue, distress), eating behavior, and physical activity, and their change in weight will covary with change in symptoms, eating behavior, and daily physical activity. Finally, it is hypothesized that participants with greater weight loss will evidence improved functioning in insulin, IL-6, IL-8, TNF-α, adiponectin, and heart rate.

ELIGIBILITY:
Phase I: Intervention Development and Refinement:

Inclusion Criteria:

* Patients:

  * Female,
  * obese (BMI >30)
  * partnered
  * diagnosis of non-metastatic breast cancer (stages I-III)
  * completed adjuvant chemotherapy and/or radiation treatment in the last 5 years
  * healthy enough to participate in a home-based walking program (if participating in intervention refinement),
  * able to speak English
  * able and willing to give informed consent.
* Partners:

  * Overweight/obese (BMI >25)
  * cohabiting partner of a woman with non-metastatic breast cancer completing adjuvant chemotherapy and/or radiation in the last 5 years
  * healthy enough to participate in a home-based walking program (if participating in intervention refinement)
  * able to speak English
  * able and willing to give informed consent.

Exclusion Criteria: for both patients and partners

* male breast cancer survivors
* non-ambulatory
* unable to provide informed consent
* have a major mental illness (i.e., schizophrenia);
* have a mental illness that is not being treated/controlled (i.e., bipolar disorder)
* reside > 100 miles from the research site.

Phase II: Feasibility, Acceptability, and Efficacy of the Intervention

Inclusion Criteria:

* Patients:

  * Female, obese (BMI >30)
  * partnered
  * diagnosis of non-metastatic breast cancer (stages I-III)
  * completed adjuvant chemotherapy and/or radiation treatment in the last 3 years
  * healthy enough to participate in a home-based walking program
  * able to speak English
  * able and willing to give informed consent.
* Partners:

  * Overweight/obese (BMI >25)
  * cohabiting partner of a woman with non-metastatic breast cancer completing adjuvant chemotherapy and/or radiation in the three years
  * healthy enough to participate in a home-based walking program
  * able to speak English
  * able and willing to give informed consent.

Exclusion Criteria: for both patients and partners

* male breast cancer survivors
* non-ambulatory
* unable to provide informed consent
* have a major mental illness (i.e., schizophrenia)
* have a mental illness that is not being treated/controlled (i.e., bipolar disorder)
* reside > 100 miles from the research site.
* Pregnant women will also be excluded from the study.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-10; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change in Weight | baseline, week 1, week 2, week 3, week 4, week 5, week 6, week 8, week 10, week 12, week 14, week 16, week 18, post-treatment (approximately 18-20 weeks), 3 months post-treatment (approximately 30-32 weeks)
  Participants will be weighed at each assessment and each session.
Change in steps per day | Through study completion (an average of 31 weeks)
  Participants will wear wireless activity trackers (Fitbits) to measure daily activity (e.g., steps taken). Participants will be provided with the activity trackers by study staff and begin to use the trackers following the pre-treatment assessment. Participants will continue to use the trackers throughout treatment. Participants will return the Fitbits to the study staff upon completion of the study.
Change in 6 minute walk ability score | baseline, post-treatment (approximately 18-20 weeks), 3 months post-treatment (approximately 30-32 weeks)
  The 6-minute walk test is a self-paced, timed test of the total distance in meters that a patient is able to walk over a six-minute period and assesses the ability to exert effort during activity.
Change in 6 minute walk pain score | baseline, post-treatment (approximately 18-20 weeks), 3 months post-treatment (approximately 30-32 weeks)
  The degree of pain experienced during the 6-minute walk test will also be assessed.
Change in Stanford Leisure-Time Activity Categorical Item (L-Cat) | baseline , post-treatment (approximately 18-20 weeks), 3 months post-treatment (approximately 30-32 weeks)
  The L-Cat is a measure of physical activity. Individuals identify which descriptive category best describes their level of activity during leisure time in the last month. Descriptive categories range from inactive to very active.
Change in Eating Behavior | baseline , post-treatment (approximately 18-20 weeks), 3 months post-treatment (approximately 30-32 weeks)
  Participants will also be asked to complete the Dietary Instrument for Nutrition Education (DINE). The DINE is a brief assessment of the amount of fat and dietary fiber in an individual's usual diet. Participants are provided with a list of food items and asked about the frequency with which they have eaten the items per week when considering the last month.
Change in The Brief Pain Inventory (BPI) | baseline , post-treatment (approximately 18-20 weeks), 3 months post-treatment (approximately 30-32 weeks)
  The BPI is a 9-item self-report measure assessing pain severity. Participants rate their pain on a scale from 0 to 10 where 0 represents "no pain" and 10 represents "pain as bad as you can imagine." Participants also rate their level of interference from pain.
Change in Promis Fatigue Scale | pre-treatment, post-treatment (approximately 18-20 weeks), 3 months post-treatment (approximately 30-32 weeks)
  The Promis Fatigue Scale is a 6-item self-report measure of fatigue in the last week
Change in Profile of Mood States (POMS) | baseline , post-treatment (approximately 18-20 weeks), 3 months post-treatment (approximately 30-32 weeks)
  The POMS will be used to assess psychological distress. Each item is rated on a scale from 0 (not at all) to 4 (extremely) as being self-descriptive for the last seven days.
Change in Physical Activity based on the International Physical Activity Questionnaire | pre-treatment, post-treatment (approximately 18-20 weeks), 3 months post-treatment (approximately 30-32 weeks)
  Participants will also complete the International Physical Activity Questionnaire (IPAQ). This seven-item questionnaire assesses the amount of time participants have spent doing moderate and vigorous physical activities in the last seven days.
Change in eating behavior using the Three Factor Eating Questionnaire | pre-treatment, post-treatment (approximately 18-20 weeks), 3 months post-treatment (approximately 30-32 weeks)
  Eating behaviors will be assessed using the Three Factor Eating Questionnaire (TFEQ). The 21-item short-form will be used for the present study. The TFEQ measures three domains of eating behavior: 1) cognitive restraint, 2) uncontrolled eating, and 3) emotional eating.

SECONDARY OUTCOMES:
Change in Fasting insulin | baseline and 3 months post-treatment (approximately 30-32 weeks)
  Fasting insulin will be examined by taking a sample of peripheral blood from participants at the baseline and post-treatment assessments.
Change in IL-6 | baseline and 3 months post-treatment (approximately 30-32 weeks)
  The pro-inflammatory cytokine IL-6 will be examined by taking a sample of peripheral blood from participants at the baseline and post-treatment assessments.
Change in IL-8 | baseline and 3 months post-treatment (approximately 30-32 weeks)
  The pro-inflammatory cytokine IL-8 will be examined by taking a sample of peripheral blood from participants at the baseline and post-treatment assessments.
Change in TNF-alpha | baseline and 3 months post-treatment (approximately 30-32 weeks)
  The pro-inflammatory cytokine TNF-alpha will be examined by taking a sample of peripheral blood from participants at the baseline and post-treatment assessments.
Change in Adiponectin | baseline and 3 months post-treatment (approximately 30-32 weeks)
  The anti-inflammatory cytokine adiponectin will be examined by taking a sample of peripheral blood from participants at the baseline and post-treatment assessments.
Change in Heart Rate | Through study completion (an average of 31 weeks)
  Heart rate will be assessed via the wireless activity trackers (Fitbit) worn by participants throughout the study.
Treatment Acceptability Questionnaire (TAQ) | post-treatment (approximately 30-32 weeks)
  The Treatment Acceptability Questionnaire (TAQ) is a six-item scale assessing whether participants view an intervention as acceptable, ethical, and effective. Items are rated on a 7-point Likert scale (e.g., 1 "very unacceptable" to 7 "very acceptable).
Change in Session attendance rate | week 1, week 2, week 3, week 4, week 5, week 6, week 8, week 10, week 12, week 14, week 16, week 18
  Treatment feasibility will be assessed by measuring the session attendance rate for each participant and each day.
Change in Use of intervention strategies | week 1, week 2, week 3, week 4, week 5, week 6, week 8, week 10, week 12, week 14, week 16, week 18
  Participants' use of intervention strategies will be assessed using a measure developed for components of the present study. Participants will be asked about how frequently treatment strategies discussed in session have been used outside of session in the past week or past month depending on the timing of the questionnaire. A scale ranging from 0 "not at all" to 5 "2 or more times a day" will be used.
Change in partner support for eating and exercise | pre-treatment, post-treatment (approximately 18-20 weeks), 3 months post-treatment (approximately 30-32 weeks)
  Partner support for eating and exercise will be assessed using a modified version of the Social Support for Diet and Exercise questionnaires. Participants will be asked to provide information about the amount of encouragement and discouragement they have received from their partner over the last three months regarding healthy eating and exercise. Items are rated on a 5 point scale from 1 "none" to 5 "very often."
Change in Self-Efficacy for Weight | pre-treatment, post-treatment (approximately 18-20 weeks), 3 months post-treatment (approximately 30-32 weeks); at each intervention session (week 1, week 2, week 3, week 4, week 5, week 6, week 8, week 10, week 12, week 14, week 16, week 18)
  The Weight Efficacy Lifestyle Questionnaire is an 8-item measure of eating self-efficacy. Participants are asked to provide information about how certain they are that they can resist overeating in difficult situation (e.g., over the weekend, when tired, etc.). Response choices range from 0= "not at all confident" to 10= "very confident."
Change in self-efficacy for managing chronic disease | pre-treatment, post-treatment (approximately 18-20 weeks), 3 months post-treatment (approximately 30-32 weeks); at each intervention session (week 1, week 2, week 3, week 4, week 5, week 6, week 8, week 10, week 12, week 14, week 16, week 18)
  The Self-Efficacy for Managing Chronic Disease Scale is a 6-item scale that asks participants to rate their confidence in doing certain activities (e.g., keep emotional distress from interfering with the things you want to do) on a scale from 1= "not at all confident" to 10= "totally confident." The wording of items was slightly altered to better match the sample intended for the present study.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline S Dorfman, PhD, Principal Investigator — Duke University
Locations (1):
- Duke Cancer Institute, Durham, North Carolina, United States